CLINICAL TRIAL: NCT07277855
Title: Evaluation of the Floor-Lift Series (FLS) Pulmonary Rehabilitation Program on Short- and Long-Term Clinical and Functional Outcomes in COPD by Program Adherence: A Single-Center Quasi-Experimental Study in a North African Setting
Brief Title: Floor-Lift Series Pulmonary Rehabilitation for COPD: Short- and Long-Term Outcomes in a North African Setting
Acronym: FLS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benazzouz Redouene Sid Ahmed (Other)
Responsible Party: Sponsor-Investigator, Benazzouz Redouene Sid Ahmed, Associate professor (maitre de conferences A) in Pneumology, Laghouat University
Organization: Laghouat University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LaghouatU
Record Dates: First submitted 2025-11-19; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Muscle Weakness | Patient
Keywords: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Floor-Lift Series; Home-Based Exercise; Equipment-Free Training; Exercise Capacity; Program Adherence; North Africa; Algeria; Culturally Adapted Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Floor-Lift Series (FLS) Program (Experimental): All participants will undergo the Floor-Lift Series (FLS) pulmonary rehabilitation program - a 9-week, progressive, equipment-free intervention combining supervised and home-based sessions. The program focuses on improving lower-limb strength, balance, and mobility through repeated floor-to-stand transitions.
  * Initial phase (Weeks 1-3): Mix of Supervised and home-based training, 7-15 repetitions/day, using wall or chair support.
  * Intermediate phase (Weeks 4-6): 15-22 repetitions/day, primarily home-based.
  * Consolidation phase (Weeks 7-9): 22 repetitions/day, independently at home. Participants receive safety instructions, telephone follow-ups for motivation, and are evaluated at baseline, week 9, and 18 months for adherence, clinical, and functional outcomes.
  Interventions: Behavioral: Floor-Lift Series (FLS) Pulmonary Rehabilitation Program

INTERVENTIONS:
Behavioral: Floor-Lift Series (FLS) Pulmonary Rehabilitation Program — A culturally adapted, low-cost, equipment-free behavioral rehabilitation program designed to enhance physical function in COPD patients with difficulty rising from the floor. The intervention involves progressive daily floor-to-stand exercises integrated into home practice and supervised sessions over nine weeks. Long-term follow-up evaluates sustained adherence and clinical benefits at 18 months.
  Other Names: FLS Program

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of morbidity and functional disability, with pulmonary rehabilitation (PR) representing one of the most effective non-pharmacological interventions. However, access to conventional PR programs remains extremely limited in many regions, particularly in North Africa, where resources, infrastructure, and patient adherence pose major challenges.

The Floor-Lift Series (FLS) program was developed as a culturally adapted, equipment-free, and low-cost PR alternative. It is based on progressive floor-to-stand transitions - movements deeply integrated into daily routines and familiar in the local cultural context - to enhance feasibility and adherence.

This prospective quasi-experimental study will evaluate both the short-term and long-term effects of the FLS program in COPD patients with baseline muscle dysfunction limiting their ability to rise from the floor. The short-term phase involves a 9-week intervention combining supervised and home-based training in three progressive stages (initial, intermediate, and consolidation). The long-term phase includes follow-up assessments at 18 months to evaluate sustained adherence and maintenance of clinical and functional improvements.

The primary outcome is the completion rate, defined as achieving ≥22 daily floor-lift repetitions during the final intervention phase and maintaining adherence at long-term follow-ups. Secondary outcomes include changes in dyspnea (mMRC), exertional effort (Borg CR10), disease impact (CAT), mobility (Timed Up and Go), flexibility (fingertip-to-floor distance), exercise capacity (6-minute walk test and 1-minute sit-to-stand test), and the composite BODE index.

Safety and psychosocial factors influencing adherence will be monitored throughout the study. The trial aims to provide evidence for a scalable, culturally relevant rehabilitation model for COPD management in resource-limited settings.

DETAILED DESCRIPTION:
This prospective, single-center, quasi-experimental longitudinal study will be conducted at the Department of Pulmonology, Ali Ben Deghine Hospital, Laghouat, Algeria. The study will include adult patients with confirmed COPD (according to GOLD 2023 criteria: post-bronchodilator FEV1/FVC <0.7 and compatible clinical symptoms such as dyspnea or chronic cough) presenting with muscle weakness or difficulty rising from the floor. Participants will be recruited consecutively during outpatient consultations and will provide written informed consent before enrollment.

Intervention Description The Floor-Lift Series (FLS) is a 9-week progressive training program designed to strengthen lower-limb and core muscles through repeated floor-to-stand transitions.

* Initial phase (Weeks 1-3): Supervised and home-based training, 7-15 repetitions/day, using wall or chair support.
* Intermediate phase (Weeks 4-6): 15-22 repetitions/day, mainly home-based practice with telephonic follow-up.
* Consolidation phase (Weeks 7-9): 22 repetitions/day, performed independently at home.

Participants are instructed on safety measures and encouraged to integrate the exercises into daily routines. Telephone follow-ups ensure adherence and detect adverse events.

Follow-up and Assessments Evaluations will be performed at baseline, after 9 weeks, and at 18 month follow-ups.

* Primary outcome: program completion (≥22 daily FLS).
* Secondary outcomes:

  * Clinical measures: mMRC, Borg CR10, CAT, and BODE index.
  * Functional performance: Timed Up-and-Go (TUG), fingertip-to-floor distance (FFD), 6-minute walk distance (6MWD), and 1-minute sit-to-stand repetitions (STS).
  * Predictors of non-completion (sociodemographic, medical, and psychosocial).
  * Long-term adherence and maintenance of benefits. Safety data, exacerbations, musculoskeletal symptoms, and motivational barriers will be systematically recorded.

Analysis Plan Data will be analyzed using R software (v4.5.1). Categorical variables will be summarized as frequencies, continuous variables as medians (IQR). Between-group comparisons (completers vs non-completers) will use Mann-Whitney or Fisher's exact tests. Within-group changes will be analyzed using Wilcoxon signed-rank tests. Long-term adherence and maintenance will be evaluated with mixed-effects models. Significance will be set at p < 0.05.

Ethics and Dissemination The study protocol has been approved by the Ethics Committee of the Faculty of Medicine, University of Laghouat (Ref. 12/2024). Participation is voluntary, and data will be anonymized. Results will be disseminated through peer-reviewed publications, national and international respiratory conferences, and open-access repositories when applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Chronic Obstructive Pulmonary Disease (COPD) according to GOLD 2023 criteria (post-bronchodilator FEV1/FVC <0.7 and compatible clinical symptoms such as dyspnea or chronic cough) .
2. Presence of muscle dysfunction limiting or complicating the ability to rise from the floor.
3. Clinically stable condition (no COPD exacerbation within the past 8 weeks).
4. Provided written informed consent.

Exclusion Criteria:

1. Acute COPD exacerbation or hospitalization within the previous 8 weeks.
2. Recent myocardial infarction, unstable angina, or decompensated heart failure.
3. Severe neurological, orthopedic, or rheumatologic condition preventing safe floor exercise.
4. Cognitive impairment interfering with understanding or cooperation.
5. Refusal or withdrawal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence rate to the Floor-Lift Series (FLS) program | At 9 weeks (end of intervention), and 18 months after program initiation.
  Adherence to the Floor-Lift Series (FLS) pulmonary rehabilitation program will be defined as meeting the target of 22 floor-to-stand transitions (FLS) per day during the consolidation phase (weeks 7-9). The primary outcome will be the proportion of participants who reach this adherence criterion at the end of the 9-week program. The same adherence criterion will be reassessed at 18 months to evaluate long-term maintenance. Higher adherence rates indicate better engagement with the program and greater feasibility of sustained implementation.

SECONDARY OUTCOMES:
Change in dyspnea severity (modified Medical Research Council Dyspnea Scale, mMRC) | Baseline, 3 weeks, 6 weeks, 9 weeks, and 18 months.
  Dyspnea will be measured using the modified Medical Research Council (mMRC) Dyspnea Scale, which ranges from 0 (no dyspnea) to 4 (very severe dyspnea). Higher scores indicate worse breathlessness and functional limitation. Change in mMRC score will be assessed from baseline to post-intervention (9 weeks) and at long-term follow-up (18 months). Negative changes (lower scores) will reflect clinical improvement, whereas positive changes (higher scores) will indicate worsening dyspnea.
Change in perceived exertion (modified Borg Category-Ratio 10 Scale, CR10) | Baseline, 3 weeks, 6 weeks, 9 weeks, and 18 months.
  Perceived exertion during daily activities and during floor-lift exercises will be rated using the modified Borg Category-Ratio 10 (CR10) Scale, which ranges from 0 ("nothing at all") to 10 ("maximal"). Higher scores indicate greater perceived exertion and worse exercise tolerance. Change in Borg CR10 score will be calculated from baseline to each follow-up assessment (9 weeks, and 18 months). Decreases in score will indicate improved tolerance to effort, while increases will reflect worsening perceived exertion.
Change in disease impact (COPD Assessment Test, CAT) | Baseline, 9 weeks, and 18 months.
  COPD-related health status will be assessed using the COPD Assessment Test (CAT), an 8-item questionnaire with total scores ranging from 0 to 40. Higher CAT scores indicate worse symptom burden and poorer health status. Change in CAT total score will be evaluated from baseline to 9-week, and 18-month assessments. Negative changes (lower scores) will indicate an improvement in COPD-related health status, whereas positive changes (higher scores) will indicate deterioration.
Change in mobility (Timed Up-and-Go test, TUG) | Baseline, 9 weeks, and 18 months.
  Mobility and functional balance will be assessed using the Timed Up-and-Go (TUG) test, reported in seconds. Participants stand up from a chair, walk 3 meters, turn, walk back, and sit down. There is no fixed upper limit for TUG time. Higher TUG times indicate worse mobility and higher fall risk, whereas lower times indicate better functional mobility. Change in TUG time will be evaluated from baseline to post-intervention and long-term follow-up.
Exercise capacity - 6-minute walk distance (6MWD) | Baseline, 9 weeks, and 18 months.
  Exercise capacity will be evaluated using the 6-Minute Walk Test (6MWT), reported as 6-minute walk distance (6MWD) in meters. Participants are instructed to walk as far as possible along a flat corridor for 6 minutes. Higher 6MWD values indicate better exercise capacity, whereas lower values indicate reduced functional capacity. Change in 6MWD will be assessed from baseline to post-intervention and long-term follow-up.
Lower-Limb Functional Strength and Endurance - 1-minute Sit-to-Stand (STS) | Baseline, 9 weeks, and 18 months.
  Lower-limb functional strength and functional capacity will be assessed using the 1-Minute Sit-to-Stand (1-min STS) test, reported as the number of complete sit-to-stand repetitions performed in 60 seconds from a standard chair without using the arms. Higher repetition counts indicate better lower-limb strength and functional capacity, whereas lower counts indicate poorer performance. Change in 1-min STS repetitions will be evaluated from baseline to post-intervention and long-term follow-up.
Trunk and Hamstring Flexibility - Fingertip-to-Floor Distance (FFD) | Baseline, 9 weeks, and 18 months.
  Flexibility of the posterior chain will be assessed using the Fingertip-to-Floor Distance (FFD), measured in centimeters during a standardized forward bend with knees extended. An FFD of 0 cm indicates that the fingertips reach the floor, reflecting better flexibility, whereas higher positive values indicate reduced flexibility (greater distance between fingertips and floor). Change in FFD will be evaluated from baseline to post-intervention and long-term follow-up; decreases in FFD indicate improved flexibility, while increases indicate worsening flexibility.
Change in composite prognosis index (BODE Index) | Baseline, 9 weeks, and 18 months.
  Overall COPD prognosis will be assessed using the BODE Index (Body mass index, Airflow Obstruction, Dyspnea, Exercise capacity). The BODE Index is a composite score ranging from 0 to 10, calculated from four components: body mass index (BMI, kg/m²), post-bronchodilator FEV₁ percent predicted, dyspnea severity measured by the modified Medical Research Council (mMRC) Dyspnea Scale (0-4), and exercise capacity measured by the 6-minute walk distance (6MWD, meters). Each component is categorized and assigned points according to the original BODE model; component points are then summed to obtain the total BODE score. Higher BODE scores indicate a worse prognosis (higher risk of mortality and hospitalizations), whereas lower scores indicate a more favorable prognosis. The primary reported value for this Outcome Measure will be the total BODE Index score and its change from baseline at 9 weeks, and 18 months.
Change in airflow obstruction (post-bronchodilator FEV₁ percent predicted) | Baseline, 9 weeks, 18 months.
  Airflow obstruction will be assessed by post-bronchodilator spirometry, reporting forced expiratory volume in 1 second (FEV₁) as percent of the predicted value for age, sex, height, and ethnicity. Lower FEV₁ percent predicted indicates more severe airflow limitation. Change in FEV₁ percent predicted will be evaluated from baseline to post-intervention (9 weeks) and at 18 months follow-up assessments; increases in FEV₁ percent predicted will indicate improvement, whereas decreases will indicate worsening obstruction.
Change in Lower-Limb Muscle Strength (Isometric 1RM Tests) | Baseline and 9 weeks and 18 months
  Isometric maximal voluntary contraction (1RM, in kilograms of force) for:
  * Knee extension
  * Knee flexion The outcome is the change in 1RM for each movement from baseline to end of program (and follow-up if repeated). Higher values indicate greater muscle strength.
Change in Upper-Limb and Pectoral Muscle Strength (Isometric 1RM Tests) | Baseline and 9 weeks and 18 months.
  Isometric maximal voluntary contraction (1RM, kgf) for:
  * Shoulder flexion
  * Pectoral press Again, outcome is change in 1RM from baseline to end of program. Higher values indicate greater strength.
Change in Muscular Endurance at 50% 1RM | Baseline and 9 weeks and 18 months.
  Muscular endurance tests at 50% of 1RM, recorded as number of repetitions or time maintained (depending on your exact protocol) for:
  * Knee extension
  * Knee flexion
  * Shoulder flexion
  * Pectoral press Outcome: change in endurance measure from baseline to end of program. Higher values = better endurance.

OTHER OUTCOMES:
Incidence of adverse events | Throughout the 9-week program and during the 18 -month follow-up period.
  Number and nature of musculoskeletal, cardiovascular, or respiratory adverse events reported during or after FLS training.

CONTACTS AND LOCATIONS:
Overall Officials: Redouene Sid Ahmed Benazzouz, DESM, Study Director — Laghouat Public Hospital; Faculty of Medicine, Laghouat University; Hanane Fatemi, MD, Principal Investigator — Laghouat Public Hospital; Faculty of Medicine, Laghouat University
Locations (1):
- Laghouat University, Laghouat, Laghouat Province, Algeria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the main publication will be shared, including baseline characteristics, intervention adherence, and all primary and secondary outcome measures (dyspnea, perceived exertion, exercise capacity tests, flexibility measures, BODE index, exacerbations, and hospitalizations). No directly identifying information will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 6 to 12 months after publication of the main trial results and for at least 5 years thereafter, or longer if scientifically justified and if resources allow.
Access Criteria: De-identified IPD will be made available to qualified researchers affiliated with academic or public institutions, for non-commercial research questions that are consistent with the objectives of the trial. Investigators must submit a written request with a brief proposal and analysis plan. Access will be granted after approval by the principal investigator and, if required, the local ethics committee, and following signature of a data use agreement specifying data security, prohibition of re-identification, and obligation to acknowledge the original study.